CLINICAL TRIAL: NCT07208305
Title: Olanzapine Plus Metoclopramide for the Prevention of Opioid-Induced Nausea and Vomiting
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Doctor, Affiliated Hospital of Qinghai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AHQU-2025003
Record Dates: First submitted 2025-09-21; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Nausea; Vomiting
Keywords: Olanzapine; Metoclopramide; Opioid; Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Olanzapine; Metoclopramide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No intervention group (No Intervention): The group did not receive conventional additional preventive treatment.
- Olanzapine plus metoclopramide group (Active Comparator): The experimental group received olanzapine (2.5mg/ night, oral, taken 30 minutes before opioid drugs on the first day of treatment) plus metoclopramide (10mg/ time, oral, 3 times a day) for 7 days.
  Interventions: Drug: Olanzapine; Drug: Metoclopramide

INTERVENTIONS:
Drug: Olanzapine — Oral olanzapine (2.5mg per night, oral, 30 minutes before taking opioids on the first day of treatment), for 7 consecutive days.
  Arms: Olanzapine plus metoclopramide group
Drug: Metoclopramide — Metoclopramide (10mg/ time, orally, 3 times a day) was taken orally for 7 days.
  Arms: Olanzapine plus metoclopramide group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of olanzapine plus metoclopramide in preventing opioid-induced nausea and vomiting (OINV) in adult patients with advanced cancer who are initiating strong opioid therapy. The main questions it aims to answer are: (1) Does the combination of olanzapine and metoclopramide reduce the incidence of OINV? (2)What adverse events do participants experience when taking the combination of olanzapine and metoclopramide? Researchers will compare the olanzapine-metoclopramide combination to a no prophylactic treatment control group to determine whether the combination is effective in preventing OINV.

Participants will: Take olanzapine (2.5 mg/day ) and metoclopramide (10 mg three times daily) or receive no prophylaxis for 7 days; Through follow-up, nausea, vomiting, the time of the first attack of nausea and vomiting, the duration of nausea and vomiting, the use of strong opioids and adverse events were evaluated and recorded, as well as the pain score (using NRS) and quality of life (EQ-5D-5L) of the patients were evaluated at baseline and on day 7.

DETAILED DESCRIPTION:
Patients were randomly assigned in a 1:1 ratio to: The study group received olanzapine 2.5mg qn+ metoclopramide 10mg tid po for a total of 7 days for preventive treatment; The control group did not receive preventive treatment. Both groups could receive other treatments recommended by doctors after the appearance of OINV.

ELIGIBILITY:
Inclusion criteria

1. Patients with malignant tumors diagnosed by pathology or histology;
2. Patients diagnosed with locally advanced or advanced stages by imaging;
3. Age: 18 to 80 years old;
4. The eastern cooperative oncology group (ECOG) performance status of 0-3;
5. The expected survival period shall be no less than 4 weeks;
6. Moderate or severe cancer pain with a Numerical Rating Scale (NRS) score of ≥ 4 points;
7. Be able to take oral medication;
8. Initial treatment with potent opioid painkillers (such as morphine, oxycodone, fentanyl, etc.);
9. No systemic chemotherapy or radiotherapy was received within one month prior to selection, and no drugs that may induce nausea and vomiting were used.
10. There were no gastrointestinal discomforts such as nausea or vomiting at the time of selection, and no intestinal obstruction.
11. Possess normal comprehension and communication skills, be capable of completing research evaluations and following research procedures.

Exclusion criteria

1. Diabetic patients with a clear diagnosis and poorly controlled blood sugar levels;
2. There are symptoms of nausea or vomiting;
3. Symptomatic intracranial diseases, such as brain metastases or leptomeningeal metastasis;
4. Received chemotherapy drug treatment within one week before the trial medication or during the trial period;
5. Receive radiotherapy for the head, abdomen or pelvic cavity within one week before the trial or during the trial;
6. New drugs with emetic or antiemetic effects have been used within 48 hours before the start of the trial;
7. Patients with severe electrolyte imbalance, abnormal kidney or liver function;
8. Patients with gastrointestinal bleeding;
9. Pregnant or lactating women;
10. Patients diagnosed with breast cancer;
11. Those whose electrocardiogram examination indicates heart disease or prolonged QTc interval;
12. There is a history of allergy or contraindications to olanzapine or metoclopramide.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with complete control (CC) in both groups during the study period (0-7 days after the initiation of opioid treatment); CC is defined as: no vomiting attack, no rescue medications are used, and no nausea. | One week
  During the 7-day study period after opioid treatment, the proportion of patients achieving CC was compared between the two groups.

SECONDARY OUTCOMES:
The proportion of patients in the two groups who achieved complete response (CR) during the study period (0-7 days after the initiation of opioid treatment); CR is defined as patients who have no vomiting/retching or rescue medications | One week
  The proportion of patients achieving overall stage complete response is defined aspatients who have no vomiting/retching or rescue medications during 0 to 7 days after the initiation of opioid treatment.
Proportion of patients adherent to strong opioid therapy during intervention period (Day 0-7) and extended follow-up (Day 8-14). | Two weeks
  Adherence will be assessed based on both daily opioid use and prescribed dose compliance. The results will be summarized as the percentage of adherent patients in each study group for Day 0-7 and Day 8-14.
The proportion of patients without nausea in both groups during the study period (0-7 days after the start of opioid treatment); | One week
  The proportion of patients without nausea in both groups during the study period (0-7 days after the start of opioid treatment); The definition of no nausea is: the visual analogue scale score = 0
The proportion of patients without vomiting in the two groups during the study period (0-7 days after the start of opioid treatment); | One week
  The proportion of patients without vomiting in the two groups during the study period (0-7 days after the start of opioid treatment);
During the study period(0-7 days after the initiation of opioid treatment), the median time differences in the first occurrence of nausea and the first occurrence of vomiting between the two groups of patients | One week
  The median time differences in the first occurrence of nausea and the first occurrence of vomiting between the two groups of patients
During the study period (0-7 days after the start of opioid treatment), the difference in the cumulative duration of nausea and vomiting attacks between the two groups of patients; | One week
  The difference in the total duration of nausea and vomiting episodes between the two treatment groups was assessed over the 7-day study period following opioid initiation. For each patient who experienced symptoms, the cumulative duration (in days) of all nausea and vomiting events was calculated based on daily diary entries and follow-up records. The mean or median of these cumulative durations was then compared between the intervention and control groups.
The differences in the proportion of patients who did not use rescue antiemetics and the cumulative use of rescue antiemetics between the two groups during the study period (0-7 days after the initiation of opioid therapy) | One week
  The need for rescue antiemetics was assessed by comparing both the proportion of patients who remained rescue-free and the mean number of rescue medication administrations per patient between the two groups during the 7-day intervention period.
The proportion of patients who achieved cancer pain relief (defined as an Numeric Rating Scale (NRS) score ≤ 3 points) from baseline to the end of the 7-day intervention. | One week
  The NRS is a validated, 11-point scale widely used for self-reporting cancer pain intensity. Patients are asked to rate their pain from 0 (representing "no pain") to 10 (representing "the worst pain imaginable").
The difference in the change of quality of life between the two groups from baseline to the end of the 7-day intervention, as assessed by the European Quality of Life 5-Dimension 5-Level Scale (EQ-5D-5L). | One week
  The quality of life will be evaluated using the EQ-5D-5L questionnaire, which is a standardized tool consisting of five dimensions (activity ability, self-care, daily activities, pain/discomfort, anxiety/depression), with each dimension having five levels. The score will be converted into a single indicator value, ranging from -0.594 to 1.000 (where 1.000 represents the full life value and a lower score indicates a poorer health status). The higher the score, the better the health condition. The main analysis will compare the average change of the EQ-5D-5L index score from baseline to day 7 between the intervention group and the control group.
Incidence of treatment-emergent adverse events related to olanzapine or metoclopramide during the 7-day study period, graded by the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0. | One week
  The safety profile of the prophylactic regimen will be assessed by comparing the proportion of patients in each group who experience at least one adverse event related to olanzapine or metoclopramide during the 7-day study period. All adverse events will be graded for severity according to the NCI CTCAE v5.0.
The difference in overall survival (OS) rates between the two groups. | Half a year
  After the study began, survival follow-up was conducted on the patients, recording the time from the start of the study to the occurrence of the event or the follow-up, as well as the survival status of the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai University Affiliated Hospital, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: Yes